CLINICAL TRIAL: NCT02654145
Title: A Multi-centre, Open Label, Single Arm, 32-week Treatment Study in Subjects With Severe Eosinophilic Asthma Not Optimally Controlled With Current Omalizumab Treatment Who Are Switched From Omalizumab to Mepolizumab 100mg Subcutaneous (Study Number 204471- the OSMO Study)
Brief Title: Omalizumab to Mepolizumab Switch Study in Severe Eosinophilic Asthma Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 204471; 2015-003697-32 (EudraCT Number)
Expanded Access: NCT00244686 (No longer available)
Record Dates: First submitted 2016-01-11; First posted 2016-01-13 (Estimated); Results first posted 2018-01-31 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Asthma
Keywords: mepolizumab; Omalizumab; SGRQ; severe eosinophilic asthma; ACQ; exacerbations
MeSH Terms: conditions — Asthma; Pulmonary Eosinophilia | interventions — mepolizumab; Albuterol; Omalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Omalizumab switch to mepolizumab 100mg SC every 4 weeks (Experimental): Subjects with severe eosinophilic asthma who are receiving omalizumab will enter a run-in period for a minimum of one week and a up to 4 weeks. Subjects will remain on their current maintenance therapy throughout the run-in period, including omalizumab. At Visit 2 (week 0) subjects will discontinue omalizumab treatment and will be switched to receiving mepolizumab 100 mg SC every 4 weeks for 28 weeks. Except for omalizumab, subjects will remain on their current maintenance therapy throughout the open-label treatment period. Albuterol/salbutamol metered dose inhalers (MDIs) will be provided as rescue medication during treatment period.
  Interventions: Drug: Mepolizumab 100mg SC; Drug: Albuterol/salbutamol MDIs; Drug: Omalizumab

INTERVENTIONS:
Drug: Mepolizumab 100mg SC — At Visit 2 (Week 0) eligible subjects will receive mepolizumab 100mg SC into the upper arm or thigh every 4 weeks over a period of 28 weeks.
Drug: Albuterol/salbutamol MDIs — Albuterol/salbutamol metered dose inhalers (MDIs) will be provided as rescue medication during treatment period.
Drug: Omalizumab — Subjects receiving omalizumab will enter in a run-in period and will continue to receive omalizumab throughout the run-in period. At Visit 2 (week 0) subjects will discontinue omalizumab.

SUMMARY:
Mepolizumab is an anti-interleukin-5 ( IL-5) monoclonal antibody that neutralizes IL-5 and reduces eosinophil counts in both sputum and blood. Omalizumab an anti-immunoglobulin E (IgE) monoclonal antibody (mAb) is effective in the treatment of moderate to severe allergic asthma. The aim of this study is to investigate whether subjects not optimally controlled on their current omalizumab treatment, who are eligible for therapy with mepolizumab can be effectively and safely switched to treatment with mepolizumab to improve asthma control. The study will provide data on the efficacy, safety, immunogenicity, and tolerability of mepolizumab when switched directly from omalizumab without any wash-out. The learnings from this study may help guide physicians when substituting one biologic with another for the treatment of patients with severe eosinophilic asthma.

The study will be a multi-centre, open-label single arm trial. Patients with severe eosinophilic asthma who are receiving omalizumab, but are not optimally controlled will be eligible to participate. Subjects will remain on their current maintenance therapy including omalizumab throughout the run-in period for a minimum of one week and up to 4 weeks. At Visit 2 (week 0) subjects will discontinue their omalizumab treatment and be switched to mepolizumab 100 mg subcutaneous (SC) every 4 weeks for 28 weeks. The treatment period is 32 weeks, including an Exit Visit/Early Withdrawal Visit, 4 weeks following the subject's last dose of mepolizumab.

ELIGIBILITY:
Inclusion Criteria:

* At least 12 years of age at the time of signing the informed consent. For those countries where local regulations permit enrolment of adults only, subject recruitment will be restricted to those who are >= 18 years of age.
* Asthma: A physician diagnosis of asthma for >=2 years that meets the National Heart and Lung Institute guidelines.
* Forced expiratory volume in 1 second (FEV1): Persistent airflow obstruction as indicated by: For subjects >=18 years of age at Visit 1, a pre-bronchodilator FEV1 <80% predicted recorded at Visit 1, For subjects 12-17 years of age at Visit 1, a pre-bronchodilator FEV1 <90% predicted recorded at Visit 1 or FEV1/ Forced Vital Capacity (FVC) ratio <0.8 recorded at Visit 1
* Eosinophilic asthma: Airway inflammation characterized as eosinophilic in nature as indicated by one of the following: A peripheral blood eosinophil count of >=300 cells/microliter (uL) that is related to asthma demonstrated in the past 12 months prior to Visit 1 or a peripheral blood eosinophil count of >=150 cells/uL at Visit 1 that is related to asthma.
* Inhaled Corticosteroid: A well-documented requirement for regular treatment with high-dose inhaled corticosteroid (ICS) in the 12 months prior to Visit 1 with or without maintenance oral corticosteroids (OCS). For 18 years of age and older: ICS dose must be >=880 microgram (ug)/day fluticasone propionate (FP) (ex-actuator) or equivalent daily. For ICS/ Long-Acting Beta-2-Agonists (LABA) combination preparations, the highest approved maintenance dose in the local country will meet this ICS criterion. For subjects 12-17 years of age at Visit 1: ICS dose must be >=440 ug/day fluticasone propionate (FP) (ex-actuator) or equivalent daily, For ICS/LABA combination preparations, the highest approved maintenance dose in the local country will meet this ICS criterion.
* Controller Medication: Current treatment with an additional controller medication, besides ICS, for at least 3 months or a documented failure in the past 12 months of an additional controller medication for at least 3 successive months. [e.g., LABA, leukotriene receptor antagonist (LTRA), or theophylline.]
* Asthma symptoms not optimally controlled: An ACQ-5 score of >=1.5 recorded at Visit 1.
* Omalizumab Treatment: Receiving omalizumab, based on weight and IgE levels, for at least the 4 months prior to Visit 1.
* Exacerbation history: Previously confirmed history of two or more exacerbations requiring treatment with systemic corticosteroids (intramuscular, intravenous, or oral) in the 12 months prior to Visit 1 despite the use of high-dose ICS. For subjects receiving omalizumab for >=8 months, at least one exacerbation must have occurred while on omalizumab treatment. For subjects receiving maintenance oral corticosteroids, the corticosteroid treatment for the exacerbations must have been a two-fold dose increase or greater.
* Male or eligible Female: Females: a) Non-reproductive potential defined as :Pre-menopausal females with one of the following: Documented tubal ligation, Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion, Hysterectomy, Documented Bilateral Oophorectomy, Postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause (refer to laboratory reference ranges for confirmatory levels)]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment. b) Reproductive potential and agrees to follow one of the options listed in the Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) from 30 days prior to the first dose of study medication and until at least five terminal half-lives or until any continuing pharmacologic effect has ended, whichever is longer, after the last dose of study medication and completion of the Exit visit/Early Withdrawal visit.The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in this protocol.

Exclusion Criteria:

* Concurrent Respiratory Disease: Presence of a known pre-existing, clinically important lung condition other than asthma. This includes current infection, bronchiectasis, pulmonary fibrosis, bronchopulmonary aspergillosis, or diagnoses of emphysema or chronic bronchitis (chronic obstructive pulmonary disease other than asthma) or a history of lung cancer.
* Malignancy: A current malignancy or previous history of cancer in remission for less than 12 months prior to screening (subjects that had localized carcinoma of the skin which was resected for cure will not be excluded).
* Liver disease: Subjects must not be enrolled in the study if :At screening (Visit 1) Alanine Transaminase (ALT) >2x Upper Limit of Normal (ULN); and bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%) Current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones or otherwise stable chronic liver disease per investigator assessment). Stable chronic liver disease should generally be defined by the absence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, oesophageal or gastric varices, or persistent jaundice, or cirrhosis.
* Hepatitis status: Diagnosis of chronic hepatitis B, as evidenced by positive Hepatitis B surface antigen (HBsAg) at Visit 1. Chronic stable hepatitis C (e.g.,positive hepatitis C antibody test result at screening (Visit 1) or within 3 months prior to first dose of study treatment) are acceptable if subject otherwise meets entry criteria.
* Cardiovascular: Subjects who have severe or clinically significant cardiovascular disease uncontrolled with standard treatment. Including but not limited to: a) known ejection fraction of <30% or b) severe heart failure meeting New York Heart Association Class IV classification or c) hospitalised in the 12 months prior to Visit 1 for severe heart failure meeting New York Heart Association Class III or d) angina diagnosed less than 3 months prior to Visit 1 or at Visit 1
* Subjects with QT interval corrected (QTc) > 450 milliseconds (msec) or QTc > 480 msec in subjects with Bundle Branch Block at screening Visit 1.The QTc is the QT interval corrected for heart rate according to Bazett's formula (QTcB), Fridericia's formula (QTcF), and/or another method, machine-read or manually over-read. The specific formula that will be used to determine eligibility and discontinuation for an individual subject should be determined prior to initiation of the study. In other words, several different formulae cannot be used to calculate the QTc for an individual subject and then the lowest QTc value used to include or discontinue the subject from the trial.For purposes of data analysis, QTcB, QTcF, another QT correction formula, or a composite of available values of QTc will be used.
* Other Concurrent Medical Conditions: Subjects who have known, pre-existing, clinically significant endocrine, autoimmune, metabolic, neurological, renal, gastrointestinal, hepatic, haematological or any other system abnormalities that are uncontrolled with standard treatment.
* Eosinophilic Diseases: Subjects with other conditions that could lead to elevated eosinophils such as Hypereosinophilic Syndromes, including Churg-Strauss Syndrome (Eosinophilic Granulomatosis with Polyangiitis [EGPA]), or Eosinophilic Esophagitis. Subjects with a known, pre-existing parasitic infestation within 6 months prior to Visit 1 are also to be excluded.
* Immunodeficiency: A known immunodeficiency (e.g., human immunodeficiency virus [HIV]), other than that explained by the use of corticosteroids taken as therapy for asthma.
* Other Monoclonal Antibodies: Subjects who have received any monoclonal antibody (other than omalizumab) to treat inflammatory disease within 5 half-lives of Visit 1.
* Smoking history: Current smokers or former smokers with a smoking history of >=10 pack years (number of pack years = (number of cigarettes per day / 20) x number of years smoked). A former smoker is defined as a subject who quit smoking at least 6 months prior to Screening Visit 1.
* Alcohol/Substance Abuse: A history (or suspected history) of alcohol misuse or substance abuse within 2 years prior to Visit 1.
* Adherence: Subjects who have known evidence of lack of adherence to controller medications and/or ability to follow physician's recommendations.
* Hypersensitivity: Subjects with allergy/intolerance to a monoclonal antibody or biologic. History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Investigator opinion: Omalizumab treatment has provided significant clinical benefit despite experiencing 2 exacerbations in the past 12 months, and potential benefit from a switch to mepolizumab would not outweigh the potential harm after omalizumab withdrawal for the subject.
* Previous participation: Previously participated in any study with mepolizumab and received investigational product (including placebo).
* Investigational Medications: Subjects who have received treatment with an investigational drug within the past 30 days or five terminal phase half-lives of the drug whichever is longer, prior to Screening (V1) (this also includes investigational formulations of marketed products).
* Pregnancy: Subjects who are pregnant or breastfeeding. Patients should not be enrolled if they plan to become pregnant during the time of study participation.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2016-03-17 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (51):
- United States (13):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Roseville, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Upland, California
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Piscataway, New Jersey
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, East Providence, Rhode Island
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Williamsburg, Virginia
- Argentina (6):
  - GSK Investigational Site, Florida, Buenos Aires
  - GSK Investigational Site, La Plata, Buenos Aires
  - GSK Investigational Site, Quilmes, Buenos Aires
  - GSK Investigational Site, San Juan Bautista, Buenos Aires
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Buenos Aires
- GSK Investigational Site, Erpent, Belgium
- Canada (8):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Sherwood Park, Alberta
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Ajax, Ontario
  - GSK Investigational Site, Mississauga, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Windsor, Ontario
  - GSK Investigational Site, Montreal, Quebec
- France (8):
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Grenoble
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Toulouse
- Germany (4):
  - GSK Investigational Site, Neu-Isenburg, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Berlin
- Netherlands (2):
  - GSK Investigational Site, Dordrecht
  - GSK Investigational Site, Rotterdam
- Spain (7):
  - GSK Investigational Site, Laredo, Cantabria
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, L'Hospitalet de Llobregat
  - GSK Investigational Site, Murcia
  - GSK Investigational Site, Pozuelo de Alarcón/Madrid
  - GSK Investigational Site, Santiago de Compostela. La Coruña.
  - GSK Investigational Site, Valencia
- Sweden (2):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/SearchAllPostings.aspx?searchparam=204471

REFERENCES:
- [Derived] Liu MC, Chipps B, Munoz X, Devouassoux G, Bergna M, Smith SG, Price RG, Galkin DV, Azmi J, Mouneimne D, Albers FC, Chapman KR. Benefit of switching to mepolizumab from omalizumab in severe eosinophilic asthma based on patient characteristics. Respir Res. 2021 May 10;22(1):144. doi: 10.1186/s12931-021-01733-9. PMID 33971856

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with severe eosinophilic asthma who were receiving omalizumab, but were not optimally controlled were enrolled in this open-label study and received mepolizumab 100 milligrams (mg) subcutaneously (SC) every 4 weeks for 32 weeks with last dose on Week 28. The study was conducted at 46 centers from 17 March 2016 to 31 May 2017.
Pre-assignment Details: Screening was performed at Visit 1 (Week -1). A total of 206 participants were screened of which 54 participants were screen failures. Seven additional participants were reported as pre-screen failures. The remaining 145 participants received at least one dose of mepolizumab.
Groups:
- Mepolizumab 100 mg SC: Eligible participants received mepolizumab 100 mg SC doses into the upper arm or thigh every 4 weeks over a period of 32 weeks, with the last dose administered at Week 28, along with their current maintenance therapy except omalizumab.
Period: Overall Study
Arm/Group | Mepolizumab 100 mg SC
Started | 145
Completed | 138
Not Completed | 7
Not completed — Lack of Efficacy | 1
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 145
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.6 (13.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86
  Male | 59
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race customized: Asian- Central/South Asian Heritage | 2
  Race customized: Asian- East Asian Heritage | 1
  Race customized: Asian- South East Asian Heritage | 2
  Race customized: Black or African American heritage | 11
  Race customized: White- Arabic/ North African Heritage | 4
  Race customized: White- White/Caucasian/European Heritage | 124
  Race customized: Multiple-Black/African American and White Heritage | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Asthma Control Questionnaire-5 (ACQ-5) Score at Week 32
Description: The ACQ-5 is a five-item, self-completed questionnaire, which is used as a measure of asthma control of a participant. The five questions (concerning nocturnal awakening, waking in the morning, activity limitation, shortness of breath and wheeze) enquire about the frequency and/or severity of symptoms over the previous week. The response options for all these questions range from zero (no impairment/limitation) to six (total impairment/ limitation) scale. ACQ-5 score range from 0 to 6. Higher scores indicates worsening of condition. Baseline was defined as the latest available assessment prior to first dose of mepolizumab. Change from Baseline at Week 32 was calculated as Week 32 value of ACQ-5 score minus Baseline value and was analyzed using Mixed Model Repeated Measures allowing for covariates of region, baseline maintenance OCS therapy, exacerbations in the year prior to the study (as ordinal variable) and visit.
Time Frame: Baseline and at Week 32
Population: Intent to treat - all participants who received at least one dose of mepolizumab
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 145
Scores on a scale | -1.45 (0.107)
Statistical Analysis 1: Comparison: Mepolizumab 100 mg SC; Test type: Superiority; p < 0.001, Mixed Model Repeated Measures — p-value is for Difference (Mepo-Placebo) calculated based on the Historical Placebo estimate of -0.55 (Standard Error: 0.05), which was estimated from a meta-analysis of studies NCT01000506 and NCT01691521 using all Placebo participants; Mean Difference (Final Values) = -0.90, 95% CI 2-sided [-1.13 to -0.66] — Difference (Mepo-Placebo) calculated based on the Historical Placebo estimate of -0.55 (Standard Error: 0.05), which was estimated from a meta-analysis of studies NCT01000506 and NCT01691521 using all Placebo participants
Statistical Analysis 2: Comparison: Mepolizumab 100 mg SC; Test type: Superiority; p < 0.001, Mixed Model Repeated Measures — p- value for Difference (Mepo-Placebo) calculated based on the Historical Placebo estimate of -0.11 (Standard Error: 0.14), which was estimated from a meta-analysis of studies NCT01691521 and NCT02281318 using Placebo participants who previously used; Mean Difference (Final Values) = -1.34, 95% CI 2-sided [-1.68 to -1.00] — Difference (Mepo-Placebo) calculated based on the Historical Placebo estimate of -0.11 (Standard Error: 0.14), which was estimated from a meta-analysis of studies NCT01691521 and NCT02281318 using Placebo participants who previously used Xolair

2. Secondary Outcome: Mean Change From Baseline in St. George's Respiratory Questionnaire (SGRQ) Score at Week 32
Description: The SGRQ Questionnaire is a well-established, self-completed tool, comprising of 50 questions with 76 weighted responses designed to measure Quality of Life in participants with diseases of airway obstruction. It consists of two parts; Part 1 produces the symptom score and Part 2 produces the activity and impact score. A Total score is also calculated which summarizes the impact of the disease on overall health status. Scores are expressed as a percentage of overall impairment where 100 represents worst possible health status and zero indicates best possible health status. Baseline was defined as the latest available assessment prior to first dose of mepolizumab. Change from Baseline at Week 32 was calculated as Week 32 value of SGRQ score minus Baseline value and was analyzed using Mixed Model Repeated Measures allowing for covariates of region, baseline maintenance OCS therapy, exacerbations in the year prior to the study (as an ordinal variable) and visit.
Time Frame: Baseline and at Week 32
Population: Intent to treat - all participants who received at least one dose of mepolizumab
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 145
Scores on a scale | -19.0 (1.64)

3. Secondary Outcome: The Rate of Clinically Significant Asthma Exacerbations Over 32 Weeks' Treatment
Description: Clinically significant exacerbations of asthma were defined as worsening of asthma which requires use of systemic corticosteroids and/or hospitalization and/or Emergency Department (ED) visits. The frequency of clinically significant asthma exacerbations over 32 weeks' treatment was analyzed using Negative Binomial Regression via generalized estimating equations with a covariate of time period (pre-treatment versus on- and off treatment).
Time Frame: Up to Week 32
Population: Intent to treat - all participants who received at least one dose of mepolizumab
Measure: Number; unit: Exacerbation rate per year
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 145
Exacerbation rate per year | 1.18
Statistical Analysis 1: Comparison: Mepolizumab 100 mg SC; Test type: Superiority; p < 0.001, Generalised Estimating Equations; Rate ratio = 0.36, 95% CI 2-sided [0.28 to 0.47] — Analysis performed using generalized estimating equation (GEE) model assuming a negative binomial distribution with a covariate of treatment period (pre-treatment , on- and off-treatment), logarithm of time as an offset variable

4. Secondary Outcome: Ratio to Baseline in Blood Eosinophil Count at Week 32
Description: Blood samples were collected at specific time points to measure blood eosinophils level for evaluation of pharmacodynamic effects in participants with a severe eosinophilic asthma phenotype when they were directly switched to mepolizumab. Baseline was defined as the latest available assessment prior to first dose of mepolizumab and ratio to Baseline at Week 32 was defined as Week 32 value divided by Baseline value and was analyzed using Mixed Model Repeated Measures allowing for covariates of region, Baseline maintenance oral corticosteroid (OCS) therapy, exacerbations in the year prior to the study (as an ordinal variable) and visit. The log transformation was applied to blood eosinophil counts prior to analysis. If a blood eosinophil count of zero was reported, it was imputed with half of the lowest possible blood eosinophil count, where applicable, prior to log transforming the data. The dispersion measure used was log standard error.
Time Frame: Baseline and at Week 32
Population: Intent to treat- all participants who received at least one dose of mepolizumab
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Mepolizumab 100 mg SC
Number analyzed (Participants) | 145
Ratio | 0.22 (0.106)

ADVERSE EVENTS:
Time Frame: The on-treatment adverse events (AEs) and on-treatment serious AEs (SAEs) are the AEs which happened on/after the first dose of mepolizumab date and before/on last dose of mepolizumab date + 28 days (up to 32 weeks).
Description: AEs and SAEs were collected in intent-To-Treat Population which comprised of all participants who received at least one dose of Mepolizumab.
Arm/Group | Mepolizumab 100 mg SC
All-Cause Mortality (participants affected / at risk) | 0/145
Serious Adverse Events (participants affected / at risk) | 16/145
Other Adverse Events (participants affected / at risk) | 107/145
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mepolizumab 100 mg SC (N=145)
Asthma (Respiratory, thoracic and mediastinal disorders) | 7 (9)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2)
Influenza (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Dental cyst (Gastrointestinal disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mepolizumab 100 mg SC (N=145)
Viral upper respiratory tract infection (Infections and infestations) | 24 (33)
Bronchitis (Infections and infestations) | 19 (23)
Influenza (Infections and infestations) | 11 (14)
Rhinitis (Infections and infestations) | 11 (11)
Sinusitis (Infections and infestations) | 8 (10)
Gastroenteritis viral (Infections and infestations) | 5 (5)
Urinary tract infection (Infections and infestations) | 5 (7)
Headache (Nervous system disorders) | 41 (89)
Dizziness (Nervous system disorders) | 5 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (20)
Back pain (Musculoskeletal and connective tissue disorders) | 13 (15)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (8)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 (7)
Neck pain (Musculoskeletal and connective tissue disorders) | 6 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (13)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 10 (12)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (15)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Fatigue (General disorders) | 14 (20)
Asthenia (General disorders) | 6 (8)
Chest pain (General disorders) | 6 (10)
Injection site reaction (General disorders) | 5 (23)
Nausea (Gastrointestinal disorders) | 11 (12)
Diarrhoea (Gastrointestinal disorders) | 9 (11)
Abdominal pain upper (Gastrointestinal disorders) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-05-08): https://cdn.clinicaltrials.gov/large-docs/45/NCT02654145/SAP_000.pdf
  • Study Protocol (2016-03-23): https://cdn.clinicaltrials.gov/large-docs/45/NCT02654145/Prot_001.pdf